CLINICAL TRIAL: NCT06616649
Title: Closed Loop Spinal Cord Stimulation for Chemotherapy Induced Peripheral Neuropathy, a Pilot Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0446; NCI-2024-08285 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SCS Implantation (Experimental): Participants will be screened on a weekly basis in the Pain Management Clinic
  Interventions: Device: Spinal cord stimulator implant

INTERVENTIONS:
Device: Spinal cord stimulator implant — Participants will receive intervention in the operating room setting

SUMMARY:
To explore the benefits of using closed loop spinal cord stimulation (SCS) in the treatment of patients experiencing painful chemotherapy induced peripheral neuropathy (CIPN) by assessing changes in pain, quality of life, pain medication use, sensory improvement through quantitative sensory testing, and improvement of gait through quantitative gait testing.

DETAILED DESCRIPTION:
Primary Objective:

To explore the impact of using closed loop spinal cord stimulation (SCS) on pain control, quality of life, and pain medication use in patients suffering from chemotherapy induced peripheral neuropathy (CIPN).

Secondary Objective:

To assess the relationship between pain control from closed loop spinal cord stimulation and any associated changes in quantitative sensory testing (QST) and quantitative gait testing (QGT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis history of CIPN of lower extremities
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of SCS
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients undergoing active chemotherapy or immunotherapy
* Patients undergoing medical litigation.
* Patients with active infection, being treated with antibiotics
* Patients that are pregnant or planning to conceive
* Patients who are receiving any investigational agents.
* Patients with brain metastases.
* Patients with cognitive impairment/psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with history of alternative forms of sensorimotor neuropathies prior to CIPN presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Through study completion; an average of 1 year
  These scales are 0-10 (0 being no pain & 10 most extreme pain).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Chung, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org